CLINICAL TRIAL: NCT01519830
Title: Significance of Iron Deficiency in Transfusion Medicine: Effects of Iron Substitution on Fatigue Und General Well Being in Healthy Blood Donors
Brief Title: Iron Substitution in Blood Donors
Acronym: ISUB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Blutspendedienst SRK Bern AG, 3008 Bern, Switzerland (Unknown); University of Bern (Other); Humanitäre Stiftung des Schweizerischen Roten Kreuzes, 3011 Bern, Switzerland (Unknown)
Responsible Party: Peter Keller, MD, Universitätklinik für Hämatologie, Inselspital Bern, CH-3010 Bern
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 010/11; Swissmedic 2011DR3145
Record Dates: First submitted 2012-01-16; First posted 2012-01-27 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Fatigue
Keywords: Anemia, Iron-Deficiency; Blood Donors
MeSH Terms: conditions — Fatigue; Anemia, Iron-Deficiency | interventions — ferric carboxymaltose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Verum (Experimental): Iron Carboxymaltose (Ferinject)
  Interventions: Drug: Iron carboxymaltose (Ferinject)
- Placebo (Placebo Comparator): 0.9% NaCl solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Iron carboxymaltose (Ferinject) — Intravenous iron
  Arms: Verum
Drug: Placebo — 0.9% NaCl solution
  Arms: Placebo

SUMMARY:
Depletion of iron stores is frequently observed in regular blood donors, but effects of iron deficiency on general health is not well studied. Recent studies in women suffering of fatigue suggest iron deficiency without concomitant anemia as a common cause of these complaints. Provided the same is true in healthy subjects, substitution of intravenous iron might result in an improvement of general well being in iron depleted blood donors.

Healthy regular blood donors will be screened for low storage iron. Qualifying subjects will be invited to participate in a randomized, placebo-controlled trial with substitution of intravenous iron or placebo (saline solution). Differences in subjectively felt fatigue and other factors of general health and well being will be assessed. If an improvement of such factors can be shown after iron replacement, relevant concerns about artificially lowering iron stores by repeated phlebotomies will arise and changes of monitoring and substitution policies in blood banking might have to be discussed.

DETAILED DESCRIPTION:
Background

Chronic iron deficiency causes anemia with impairment of physical and mental capacity. Since iron plays an essential role in many enzymes apart from oxygen carriage, iron deficiency was proposed as an independent factor impairing wellbeing also without anemia. Symptoms like fatigue, asthenia, physical weakness, mental impairment and many others have been associated with iron deficiency. Recent clinical trials with iron substitution in iron deficient women suffering of general fatigue support this hypothesis, but data are still conflicting and debated.

Low body iron stores are frequently observed in blood donors. Repeated phlebotomies may induce or aggravate severe iron deficiency. Astonishingly, little is known about the long term effects of reduced iron stores on general health of regular blood donors. Serious health impairment cannot be excluded conclusively. Since many symptoms associated with iron deficiency are subtle, they might be missed by otherwise healthy subjects.

Blood donors with borderline or decreased iron stores (i.e. serum ferritin below 50 microg/l) will be invited to participate in a randomized, placebo-controlled intervention study comparing intravenous iron carboxymaltose and a physiological saline solution (placebo). Subjectively felt fatigue, measured on a numeric rating scale from 1 to 10 as the major end point will be assessed before and six months after application of the study drug. As additional factors, various aspects of general wellbeing will be assessed using four psychometric questionnaires. Statistical analysis will compare the results before and after application of the study drug and the results of the two study arms.

Objective

1. Assessment of severity of iron deficiency in a large group of blood donors.
2. Demonstration of an improvement of fatigue after substitution of iron compared with placebo in iron deficient blood donors
3. Detection of improved general wellbeing in otherwise healthy blood donors after substitution of intravenous iron
4. Assessment of tolerability of intravenous iron in healthy blood donors

Methods

Randomized, placebo controlled interventional trial comparing the effect of intravenous iron or placebo on fatigue and various other factors of general wellbeing. Endpoints assessed on a numeric rating scale from 1 to 10 and four psychometric questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Serum-Ferritin 50 microg/l
* Eligibility for blood donation
* At least one prior blood donation

Exclusion Criteria

* Anemia
* Known intolerability of intravenous iron
* History of anaphylactic reactions
* Active systemic infections
* Signs of chronic bleeding
* Known iron overload
* Lactation
* Pregnancy
* Any disease associated with increased fatigue
* Medication associated with increased fatigue

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Difference of fatigue on a 10 point numeric scale after intravenous substitution of iron or placebo | 6 weeks
  measured by questionnaire

SECONDARY OUTCOMES:
Change of fatigue after intravenous substitution of iron | 6 weeks
  measured by questionnaire
Improvement of general wellbeing | 6 weeks
  measured by questionnaire
Number of patients with adverse events of different grades | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Peter Keller, MD, Study Chair — Department of Hematology, Bern University Hospital, Switzerland; Bernhard Lämmle, MD, Prof., Study Chair — Department of Hematology, Bern University Hospital, Switzerland; Stefano Fontana, MD, Study Chair — Blutspendedienst SRK Bern AG, Bern, Switzerland; Peter Jüni, MD, Prof., Study Chair — Institut für Sozial- und Präventivmedizin, Universität Bern, Switzerland; Roland von Känel, MD, Prof., Study Chair — Kompetenzbereich für Psychosomatische Medizin, University Hospital Bern
Locations (1):
- Department of Hematology, Bern University Hospital, Bern, Canton of Bern, Switzerland